CLINICAL TRIAL: NCT05333172
Title: The Effect Of Balance Training With Dual Task On Cognitive Status And Functionality In Elderly
Acronym: geriatric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tuğçe Poyraz İşleyen, research assistant, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10840098-604.01.01-E.7685
Record Dates: First submitted 2022-04-12; First posted 2022-04-18 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Balance; Cognitive Functions; Dual Task; Functionality; Geriatrics

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- balance exercise group (Active Comparator): The balance program was performed on soft and hard surface. Firstly the participants started the exercises on hard ground while standing. Postural balance program consisted of static and dynamic functional balance exercises (hıp flexion, hıp abduciton, semitandem stance, one leg stance, toe tips lifting). Afterwards exercises were performed on soft surface. Three sets of eight to ten repetitions of each exercise in a slow, controlled manner were performed. This section was completed 30 minitues.
  Interventions: Other: Dual task exercises
- Dual task exercises (Experimental): Dual task exercises are in two forms as motor dual task and cognitive dual task. In this study we used cognitive secondary task exercises. In addition to the exercises applied by the balance exercise group, a cognitive task was added. Participants in this group tried to count 4, 5 and 7 back from 100 while practicing balance exercises.
  The balance program was performed on soft and hard surface. Firstly the participants started the exercises on hard ground while standing. Postural balance program consisted of static and dynamic functional balance exercises (hıp flexion, hıp abduciton, semitandem stance, one leg stance, toe tips lifting). Afterwards exercises were performed on soft surface. Three sets of eight to ten repetitions of each exercise in a slow, controlled manner were performed. This section was completed 30 minitues.
  Interventions: Other: Dual task exercises

INTERVENTIONS:
Other: Dual task exercises — Dual tasks, often also referred to as secondary tasks, present an objective-direct measurement in which two tasks are to be performed simultaneously to observe performance drops in either task.
  Other Names: balance exercise group

SUMMARY:
Aging is a dynamic process that affects motor and cognitive functions. Activities of daily living and functionality, including dual task performance, are also negatively affected by these functions. The purpose of this study is to determine of balance training with dual task on cognitive function and functionality.

DETAILED DESCRIPTION:
While physiological changes occur at the level of cells, tissues and systems with aging, these changes are reflected in motor and cognitive functions. The decrease in motor functions can be cause as balance and fall problems, which are the most serious and frequently encountered problems among the elderly. Especially the fall is one of the main reasons causing the elderly to be hospitalized in the hospital and nursing home.

Balance system is one of the most affected by aging process. The balance is maintained by receiving input from several systems, for this reason it is the system that is easily and primarily affected by changes in any of these inputs. Balance disorders have been shown to be risk factor for falling in elderly. Studies have shown that balance training has been observed to improve postural control, so it is especially recommended for to reduce risk and rate of falls in the elderly.

While general cognitive capacity decreases with aging, information processing, use and recall performance is lower than younger. Therefore, elderly have difficulty in tasks that require the use of more than one information at same time.

In daily life, a motor function is often accompanied by another task. Dual task performance is a secondary motor or cognitive task that must be implemented during a main task. Therefore, ın order for the exercises to be functional, it is not enough to be focused only on motor skills, besides adding a motor or cognitive dual task is more effective than exercise alone.

The changes in neuromusculoskeletal and movement-related functions during the aging process causes a decrease in functional ability. Most daily activities require the management of motor-cognitive tasks while simultaneously processing external information. The ability to perform in daily life activities decline in elderly.

Investigators hypothesized that balance exercises with dual task would show greater significant improvements functionality and cognitive improvements than the balance exercises only.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 65-85
* Being able to communicate
* Able to walk without mobility aids
* Be volunteer for intervention

Exclusion Criteria:

* Cognitive impairment (<17 point on the Minimal Mental State Examination )
* In physiotherapy treatment that trains balance
* Balance impairment (< 20 point on the berg balance test)
* having an orthopedic problem that may affect balance performance

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
The Mini-Mental Status Examination (MMSE) | 7 minutes
  Cognitive Functioning Test
The Functional Independence Measure (FIM) | 10 minutes
  Functionality Test

SECONDARY OUTCOMES:
The Berg Balance Scale (BBS) | 5 minutes
  Balance Test
The "Timed Up and Go" test (TUG) | 3 minutes
  Physical function test
Timed sit to stand test (TSST) | 2 minutes
  Physical function test
Ten meters walk test (TMTWT) | 3 minutes
  Physical function test
Tinetti Performance Oriented Mobility Assessment(POMA) | 15 minutes
  task-oriented test that measures an older adult's gait and balance abilities.
The Montreal Cognitive Assessment (MoCA) | 10 minutes
  Cognitive Function Assesment

CONTACTS AND LOCATIONS:
Locations (1):
- Tuğçe Poyraz Işleyen, Istanbul, Turkey (Türkiye)